CLINICAL TRIAL: NCT00990769
Title: The Effect of Depth of Anesthesia as Measured by Bispectral Index (BIS) on Emergence Agitation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Heather Frederick, Dr. Heather Frederick, Duke University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Pro00015531
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Emergence Agitation
Keywords: Emergence delirium; Bispectral Index; Depth of anesthesia
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-normal BIS ("Lighter" anesthesia) (Experimental): Depth of anesthesia is titrated to a BIS of 55-60
  Interventions: Other: Depth of anesthesia
- Low-normal BIS ("Deeper" anesthesia) (Experimental): Depth of anesthesia is maintained at a BIS level of 40-45
  Interventions: Other: Depth of anesthesia

INTERVENTIONS:
Other: Depth of anesthesia — The intervention in this study is the titration of the depth of anesthesia according to the BIS monitor, as maintained by a combination of routine anesthetic agents (nitrous oxide, sevoflurane, and fentanyl).

SUMMARY:
The purpose of this study is to determine whether depth of anesthesia has an effect on emergence agitation (EA) in children age 2 - 8 years old. EA is a common problem in pediatric patients who receive general anesthesia with inhaled anesthetics, and the effect of depth of anesthesia on EA has not been studied. The study will randomize 40 children undergoing ophthalmologic surgery under general anesthesia to either light anesthesia (BIS 55-60) or deep anesthesia (BIS 40-45). EA will be measured by the peak Pediatric Assessment of Emergence Delirium (PAED) score in the recovery room, which rates agitation behaviors on a scale of 0 - 20. The hypothesis is that light anesthesia is associated with more EA.

ELIGIBILITY:
Inclusion Criteria:

* Children age 2 - 8 (inclusive) undergoing ophthalmologic surgery
* American Society of Anesthesiology (ASA) physical status 1 or 2

Exclusion Criteria:

* Surgery precluding placement of BIS monitor
* Non-English speaking, until additional language consent forms are approved
* Previous history of severe emergence agitation

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Frederick, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center - Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents or guardians of children undergoing ophthalmologic surgery were approached, when possible, at their pre-anesthesia evaluation visit. All eligible patients were notified about the study through fliers at their pre-operative visit, and eligible patients who were missed pre-operatively were approached for consent on the day of surgery.
Pre-assignment Details: Fifty-seven patients were approached for participation; of these, fourteen declined and three were unable to participate due to surgery cancellation or rescheduling.
Groups:
- High-normal BIS: Depth of anesthesia is titrated to a BIS level of 55-60
- Low-normal BIS: Depth of anesthesia is titrated to a BIS level of 40-45
Period: Overall Study
Arm/Group | High-normal BIS | Low-normal BIS
Started | 22 (Signed consent and assigned to High-normal BIS) | 18 (Signed consent and assigned to Low-normal BIS)
Completed | 22 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-normal BIS | Low-normal BIS | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 18 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.1 (2.3) | 4.3 (1.4) | 4.7 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Peak Pediatric Assessment of Emergence Delirium (PAED) Score Within the First 30 Minutes of Reaching the Recovery Room (Post-Anesthesia Care Unit)
Description: The PAED scale is a validated observational measure of five aspects of child behavior on emergence from anesthesia (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to arrive at a total score ranging from 0 - 20, with higher scores indicating greater severity of emergence agitation.
Time Frame: Within 30 minutes of arrival in recovery room
Population: All patients in each group were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-normal BIS | Low-normal BIS
Number analyzed (Participants) | 22 | 18
units on a scale | 8.6 (5.3) | 6.7 (4.6)
Statistical Analysis 1: Comparison: High-normal BIS vs Low-normal BIS; Sample size calculation concluded that 20 patients in each group would have 80% power to detect a mean difference of 4 ± 4 with alpha equal to 0.05, as would be determined by a two-sample T test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.9, Standard Deviation 5

2. Secondary Outcome: Time to Emergence From Anesthesia
Description: The time from cessation of anesthesia delivery (Sevoflurane turned off) to extubation.
Time Frame: After the completion of surgery
Population: All patients were analyzed
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | High-normal BIS | Low-normal BIS
Number analyzed (Participants) | 22 | 18
minutes | 14 (5) | 12 (4)

3. Secondary Outcome: Pain Score: Faces, Legs, Activity, Cry, and Consolability (FLACC)
Description: Pain was assessed with the Faces, Legs, Activity, Cry, and Consolability (FLACC) scale. The FLACC scale is an observational measure of child behavior in response to postoperative pain. Five subscales are rated from 0-2 on severity: facial expression, leg position and motion, psychomotor agitation, crying, and inconsolability. Subscale scores are summed to compute a total score ranging from 0-10, with 10 representing the most severe pain. In the post-operative setting, the FLACC scale is validated for cognitively intact children up to age 7 years, and was used for all children in the study.
Time Frame: Within 30 minutes of arrival in recovery room
Population: All patients were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-normal BIS | Low-normal BIS
Number analyzed (Participants) | 22 | 18
units on a scale | 5.3 (3.3) | 3.5 (3.8)

ADVERSE EVENTS:
Arm/Group | High-normal BIS | Low-normal BIS
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No